CLINICAL TRIAL: NCT05057507
Title: Realistic Computational Electrophysiology Simulations for the Targetted Treatment of Atrial Fibrillation
Acronym: ReCETT-AF
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: AC20151
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial fibrillation patients undergoing radiofrequency catheter ablation: Up to 115 patients undergoing radiofrequency catheter ablation will be enrolled.
  Interventions: Diagnostic Test: Atrial cardiac magnetic resonance imaging; Diagnostic Test: Atrial electro-anatomic mapping; Other: Atrial fibrillation symptom questionnaire; Diagnostic Test: Patch-based 2 week ambulatory monitor

INTERVENTIONS:
Diagnostic Test: Atrial cardiac magnetic resonance imaging — To include assessment of atrial size, shape, function, fibrosis and fat
Diagnostic Test: Atrial electro-anatomic mapping — To include assessment of atrial voltage and local activation time
Other: Atrial fibrillation symptom questionnaire — To include assessment of atrial fibrillation symptoms and quality of life
Diagnostic Test: Patch-based 2 week ambulatory monitor — To assess atrial fibrillation burden post-ablation

SUMMARY:
The aim of this research is to classify patients by the dominant mechanism of continuous atrial electrical activation during atrial fibrillation. This approach seeks to improve on existing classifications which are based solely on the duration of the arrhythmia (<7 days, >7 days and >1 year). This is a cohort study. Patients undergoing clinically indicated electrophysiology study or AF ablation will have invasive assessment of cardiac electrophysiological profile at the time of their planned procedure, undergo 2-week ambulatory monitoring before and after the procedure, complete symptom questionnaires before and after their procedure and undergo atrial cardiac magnetic resonance imaging before their procedure.

DETAILED DESCRIPTION:
Atrial fibrillation is a common condition causing an irregular heartbeat, breathlessness and tiredness. Atrial fibrillation occurs owing to abnormalities in the electrical circuits controlling the upper heart chambers. Atrial fibrillation can be treated with a keyhole procedure called ablation. During ablation small areas in the heart are burnt away to stop the abnormal circuits causing atrial fibrillation. Unfortunately, ablation only works for 50-90% of people. We are not sure why, but possibly because the electrical circuits responsible are different in every heart. This research will examine how these electrical circuits can be identified and treated. A new system using computer modelling will be developed to identify the electrical circuits present. In the future we hope this approach could be used to design tailor-made treatments for each patient. A combination of computer studies and studies involving patients will be used to test this new approach in this study. For this study patients who are already planned to undergo an ablation procedure will be recruited providing data for three Work Packages. Consent will be sought to access routine investigations and data for research purposes (e.g. ECGs, blood tests, ambulatory monitoring, cardiac imaging, and outpatient clinical assessment); and collect extra data for research including additional cardiac imaging, a 2-week heart monitor pre- and post-ablation, and extra electrical measurements made during the ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal atrial fibrillation or persistent atrial fibrillation diagnosed - within 24 months preceding the consent date.
* Planned radiofrequency ablation for atrial fibrillation consisting of pulmonary vein isolation.
* Able and willing to comply with study follow-up requirements
* Able and willing to provide written informed consent

Exclusion Criteria:

* Any clinical contra-indication to ablation
* Any disease limiting life expectancy to < 1year
* Contra-indication to MRI including renal dysfunction (eGFR<30ml/min)
* Potential participant currently pregnant or breast feeding
* Prior ablation, cardiac surgery or presence of any prosthetic valves
* Myocardial infarction or percutaneous coronary intervention within 3 months preceding consent date
* Hypertrophic cardiomyopathy or other inherited cardiac condition
* Presence / likely implant of any pacemaker, cardiac resynchronization therapy device or implantable defibrillator within 1 year
* Enrolment in an existing interventional atrial fibrillation study which alters treatment or follow-up.
* Use of amiodarone for any indication within 6 months prior to the planned ablation procedure
* Use of any anti-arrhythmic drug for an arrhythmia indication other than atrial fibrillation
* Prior documented cavotricuspid isthmus dependent right atrial flutter and planned cavotricuspid isthmus ablation to be performed at the time of atrial fibrillation ablation
* Unable to understand verbal or written explanations given in English or German as appropriate.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to 115 patients undergoing electrophysiological assessment will be recruited with inclusion and exclusion criteria as indicated above.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with each mechanism of atrial fibrillation defined by computational modelling | 4 years
  The primary outcome is the creation of patient specific computational models for the investigation of atrial fibrillation mechanisms in patients. Mechanisms of atrial fibrillation will be defined based on computational modelling results and each patient will be assigned to the dominant mechanism of atrial fibrillation present.

SECONDARY OUTCOMES:
Atrial properties - atrial structural and functional properties will be compared between patients in each mechanistic atrial fibrillation group (as defined in Outcome 1) | 4 years
  The secondary outcome (1) is to determine which atrial properties are associated with each mechanism of atrial fibrillation in patients. Atrial structural and functional properties will be measured using atrial magnetic resonance imaging and invasive atrial electrophysiology; and quantified as follows: Atrial structure - volume (ml), sphericity (%); fibrosis burden (%); pericardial fat volume (ml); Atrial function - conduction velocity (m/s); refractoriness (ms); atrial electrical area (cm).
Treatment effects - burden of atrial fibrillation in patients classified as 'successfully treated' compared to those classified as 'not successfully treated' using the modelling framework (as defined in Outcome 1) | 4 years
  The secondary outcome (2) is to determine how atrial properties can be modified using currently-available therapies to improve treatment for atrial fibrillation. Computer simulations will be performed in which the critical atrial properties (as defined in Outcome 2) are modified and actual treatment response will be compared to predicted treatment response by (A) correlating actual atrial fibrillation burden (% time in atrial fibrillation) with predicted atrial fibrillation burden (% time in atrial fibrillation) and (B) calculating diagnostic accuracy metrics (sensitivity, specificity, C-statistic) for prediction of atrial fibrillation inducibility and recurrence following ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D O'Neill, FRCP, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Neil Grubb, FRCP, Principal Investigator — NHS Lothian, Edinburgh; Andreas Rillig, MD, Principal Investigator — University Heart and Vascular Center, Hamburg
Locations (2):
- United Kingdom (2):
  - NHS Lothian, Edinburgh
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No